CLINICAL TRIAL: NCT00288834
Title: Outcomes of Swallowing Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Canterbury (Other)
Collaborators: University of Toronto (Other); Tan Tock Seng Hospital (Other); Fremantle Hospital and Health Service (Other); Austin Hospital, Melbourne Australia (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSF NA 4992; NZ CMRF 01/10
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2006-02

CONDITIONS: Stroke; Cerebrovascular Accident; Dysphagia
Keywords: stroke; dysphagia; rehabilitation; biofeedback
MeSH Terms: conditions — Stroke; Deglutition Disorders

INTERVENTIONS:
Behavioral: dysphagia rehabilitation

SUMMARY:
This project proposes to evaluate the relative effectiveness of four therapy protocols for pharyngeal phase swallowing impairment in the stroke population. Data derived from this study should contribute significantly to our understanding of the rehabilitative process in the neurogenic dysphagic population and will provide the foundation for the establishment of efficacious, cost-efficient patient services.

1. Research Question to be addressed

1. The utilization of SEMG biofeedback monitoring in dysphagia rehabilitation facilitates more rapid and complete recovery than traditional rehabilitation using the same swallowing exercises without exteroceptive feedback.
2. Swallowing rehabilitation provided in an intensive rehabilitative programme (10 hrs of treatment in the 1st week) facilitates more rapid and complete recovery than traditionally scheduled swallowing rehabilitation (twice weekly).

DETAILED DESCRIPTION:
This multi-site, multi-national project will evaluate the relative effectiveness of four therapy protocols for pharyngeal phase swallowing impairment in the stroke population. For this study, patients with chronic dysphagia secondary to stroke will be assigned to one of four treatment protocols. These four protocols differ in respect to the intensity of treatment and the inclusion of surface electromyography (SEMG) biofeedback as an adjunct to treatment. All patients will complete a total of 30 hours of therapy with data collection to assess progress at intervals of every 10 sessions. Treatment outcomes will be measured using a combination of physiologic and behavioral measures. Data derived from this study should contribute significantly to our understanding of the rehabilitative process in the neurogenic dysphagic population and will provide the foundation for the establishment of efficacious, cost-efficient patient services.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will represent the diagnostic categories of single event brain stem injury, right cortical stroke and left cortical stroke.
* Chronic dysphagia at least 6 months post onset secondary to single neurological event, brain stem, right cortical or left cortical stroke confirmed with CT or MRI
* Diagnosis of chronic pharyngeal phase dysphagia based on clinical and videofluoroscopic evaluation completed within 3 weeks of beginning treatment.
* Must be at least 12 months post onset with no substantial recovery of swallowing function. If patients have received prior swallowing treatment, they must be at least three months post the termination of direct treatment.
* Mini Mental Status Exam score >21

Exclusion Criteria:

* history of pre-existing dysphagia or neurologic disease prior to the onset of the current disorder.
* MMSE score < 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2006-07

PRIMARY OUTCOMES:
The following outcomes measures will be assessed after 10. 20 and 30 therapeutic sessions:
Severity rankings of swallowing pathophysiology based on videofluoroscopic swallowing studies Videofluoroscopic swallowing studies
Functional outcome ratings of associated clinical parameters (respiratory, neurological status, self help, cognitive)
Quality of life ratings (SwalQOL) In addition, quality of life ratings (SwalQOL) will be assessed at one follow-up assessment six months post discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie-Lee Huckabee, Ph.D., Principal Investigator — University of Canterbury, Van der Veer Institute for Parkinson's and Brain Research, Christchurch New Zealand; Catriona M. Steele, Ph.D., Principal Investigator — Toronto Rehabilitation Institute, Toronto Canada; Pascal van Lieshout, Ph.D., Principal Investigator — University of Toronto, Toronto Canada
Locations (9):
- Australia (2):
  - Austin and Repatriation Medical Centre, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Canada (5):
  - Glenrose Rehabilitation Centre, Edmonton, Alberta
  - Deer Lodge Centre, Winnipeg, Manitoba
  - Leonard Miller Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Trillium Health Centre, Mississauga, Ontario
- Princess Margaret Hospital, Christchurch, New Zealand
- Tan Tock Seng Hospital, Singapore, Singapore